CLINICAL TRIAL: NCT07355751
Title: The Effect of Acupuncture Treatment on Cognitive Functions and Brain Networks for Long COVID: a Multimodal Magnetic Resonance Imaging Study
Brief Title: The Effect of Acupuncture Treatment on Cognitive Functions and Brain Networks for Long COVID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tingting Luo (Other)
Responsible Party: Sponsor-Investigator, Tingting Luo, Doctor, Chengdu University of Traditional Chinese Medicine
Organization: Chengdu University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025KL-086
Record Dates: First submitted 2026-01-02; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Long Covid
Keywords: Long COVID; cognitive function; acupuncture; neuropsychological test; brain network; magnetic resonance imaging; multimodal methods
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: data analysts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verum Acupuncture group (Experimental): Acupoints with acupuncture treatment
  Interventions: Other: Acupuncture
- Sham acupuncture group (Sham Comparator): Non-acupoints with sham acupuncture treatment
  Interventions: Other: Sham acupuncture
- Waitlist control group (No Intervention): Acupoints with acupuncture treatment after 8-week waiting period

INTERVENTIONS:
Other: Acupuncture — Two sets of acupoints will be alternatively acupunctured. The first set of acupuncture points incudes Baihui (GV20), Shenting (GV24), bilateral Neiguan (PC6), Qihai (CV6), Guanyuan (CV4), bilateral Zusanli (ST36), bilateral Sanyinjiao (SP6). The second set of acupoints consist of Sishenchong (EX-HN1), bilateral Ganshu (BL18), bilateral Pishu (BL20), bilaetral Shenshu (BL23). The treatment consists of 24 sessions of 30 minutes, given within eight weeks (three sessions per week).A set of acupoints will be acupunctured each treatment session.
  Arms: Verum Acupuncture group
Other: Sham acupuncture — Nonpenetrating acupuncture on non-acupoints will be performed using Park sham acupuncture device (0.25 mm in diameter and 40 mm in length, Hwatuo, Suzhou, China) for participants. Two sets of non-acupoints will be alternatively acupunctured. The first set of sham acupoints includes bilateral non-acupoint 1, non-acupoint 2, non-acupoint 3, bilateral non-acupoint 4, bilateral non-acupoint 5. The second set consists of bilateral non-acupoint 6, bilateral non-acupoint 7, bilateral non-acupoint 8. The treatment consists of 24 sessions of 30 minutes, given within eight weeks (three sessions per week). A set of non-acupoints will be acupunctured each treatment session.
  Arms: Sham acupuncture group

SUMMARY:
Background of study:

Long COVID(LC) is a prevalent sequalae of SARS-CoV-2 infection and can affect multiple organ systems. Cognitive dysfunction is one of the most common symptoms in LC with 22% prevalence. It can persist for years and significantly reduce patients' quality of life. Brain network is the neural basis underlying human cognitive processes. Diffusion tensor imaging (DTI) and functional magnetic resonance imaging(fMRI) research has revealed that alterations of network characteristics were associated with cognitive impairments across attention, memory, executive function and language in LC. Currently, there is no accepted therapy for cognitive impairment in LC. Acupuncture, as a Traditional Chinese Medicine therapy, has potential to improve cognitive deficits for LC. However, research focusing on the impact of acupuncture on cognitive functions in LC is rare. Additionally, no one has evaluated the mechanism of acupuncture improving cognitive functions in LC.

Objective of the study:

This study aims to assess the effect of acupuncture treatment on cognitive function and explore the central mechanism of acupuncture therapy in improving cognitive function for LC using cognitive assessments, DTI and resting-state fMRI.

Study design:

A prospective, three-armed, randomized controlled trial with DTI and rs-fMRI. Adults with LC will be randomly assigned to acupuncture, sham acupuncture, or waitlist control group in a 1:1:1 ratio, receiving 8-week intervention or waiting. Cognitive function and topological attributes of brain networks will be examined at baseline and 8th week.

Study population:

Patients fulfilling World Health Organization (WHO) criteria for LC will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Fulfilling WHO criteria for long COVID
* History of confirmed COVID-19 through RT-PCR of nasopharyngeal swab or antigen test of nasal swab ;
* Having subjective cognitive problems
* Native Chinese speakers
* Right handedness
* Voluntary to participate in the study and signing the informed consent form.

Exclusion Criteria:

* Preexisting cognitive symptoms before COVID-19
* Previous or current diagnosis of chronic conditions that may affect cognitive performances (such as neurological, psychiatric disorders, organ failure, chronic infectious diseases)
* Prior loss of consciousness
* History of major surgery within a year
* Long-term use of drugs that may influence cognition(such as tranquilizer, antidepressant, immunosuppressor)
* Previous acupuncture treatment within 3 months
* Involvement of other clinical study within 4 weeks
* Obesity(BMI≥28)
* Sensory disorders(deafness, color blindness)
* Limb dysfunction
* Metal implantation
* Claustrophobia
* Pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change of Addenbrooke's Cognitive Examination-III total score from baseline to the end of 8 weeks | Baseline and 8 weeks
  Addenbrooke's Cognitive Examination-III is a cognitive screening tool, and the total score assess general cognitive function. The total score ranges from 0 to 100. Higher score indicates better general cognitive function
Change of Phonemic Fluency Test score from baseline to the end of 8 weeks | Baseline and 8 weeks
  Phonemic fluency test measures the number of correct words produced under restricted search conditions of phonemic(letter F) . Higher score indicates better language.

SECONDARY OUTCOMES:
Changes of Digit Span Test scores from baseline to the end of 8 weeks | Baseline and 8 weeks
  Digit Span Test consists of forward and backward subtests, that respectively assess attention and executive function through measuring the number of correct digit sequences. The minimum score is 0 , and the maximum scores are respectively 10 and 9 for forward and backward subtests. Higher scores indicate better attention and executive function.
Change of Symbol Digit Modality Test score from baseline to the end of 8 weeks | Baseline and 8 weeks
  Symbol Digit Modality Test assesses attention through measuring the number of correct responses within 90 seconds. The minimum score is 0, and the maximum score is 110. Higher score indicates better attention.
Changes of Trail Making Test scores from baseline to the end of 8 weeks | Baseline and 8 weeks
  Trail Making Test includes Part A(TMT-A) and Part B(TMT-B), that respectively evaluates attention and executive function via measuring the time in seconds required for completing each part of the test. Higher scores indicate worse attention and executive function.
Changes of Rey Auditory Verbal Learning Test scores from baseline to the end of 8 weeks | Baseline and 8 weeks
  Rey Auditory Verbal Learning Test evaluates different aspects of verbal memory through measuring total learning, repetitions, delayed recall, retroactive interference, and proactive interference. Higher scores for total learning and delayed recall indicate better memory, while higher scores for repetitions, retroactive interference, and proactive interference indicate worse memory.
Changes of Rey-Osterrieth Complex Figure Test scores from baseline to the end of 8 weeks | Baseline and 8 weeks
  Rey-Osterrieth Complex Figure Test evaluates visuospatial construction ability through measuring the accuracy of copy, and evaluates visual memory via measuring the accuracies of immediate and delayed recalls. Higher scores indicate better visuospatial construction and visual memory.
Changes of Stroop Test scores from baseline to the end of 8 weeks | Baseline and 8 weeks
  Stroop test consists of Stroop word test(Part A), Stroop color test(Part B) and Stroop color word test(Part C), that assess executive function through measuring the time in second required to complete each part and the number of errors for each part. Higher score for each part indicates worse executive function.
Change of Category Fluency Test Score from baseline to the end of 8 weeks. | Baseline and 8 weeks
  Category Fluency Test assesses language through measuring the number of correct words produced under restricted search condition of category(animals). Higher score for each subtest indicates better language.
Change of Action Fluency Test Score from baseline to the end of 8 weeks | Baseline and 8 weeks
  Action Fluency Test evaluates language via measures the number of correct words produced under restricted search condition of action(kitchen actions). Higher score for each subtest indicates better language
Change of Boston Naming Test score from baseline to the end of 8 weeks | Baseline and 8 weeks
  Boston Naming Test includes 30 items and evaluates language through measuring the total of correct responses. The minimum score is 0, and the maximum score is 30. Higher score indicates better language.
Change in Fatigue Severity Scale score from baseline to the end of 8 weeks | Baseline and 8 weeks
  Fatigue Severity Scale is a self-report questionnaire consisting of 9 items which are devised to evaluate the impact of fatigue on daily functioning, severity of fatigue. The minimum score is 9,and the maximum score is 63. Higher score indicate greater severity of fatigue and impact of fatigue on daily functioning.
Change of the Generalized Anxiety Disorde-7 score from baseline to the end of 8 weeks | Baseline and 8 weeks
  Generalized Anxiety Disorde-7 is a self-report questionnaire with 7 items, that assesses the level of anxiety in the past two week. The minimum score is 0, and the maximum score is 21. Higher score indicates greater severity of anxiety.
Change of Hamilton Depression Scale score from baseline to the end of 8 weeks | Baseline and 8 weeks
  Hamilton Depression Scale is the most commonly used instrument for the assessment of depression in clinical practice. It includes 24 items and assesses the level of depression through measuring factors of Anxiety/Somatization, Weight, Cognitive Impairment, Diurnal Variation, Retardation, Sleep Disturbance, and Hopelessness. The total score range is 0 to 76. Higher total score indicates greater level of depression.
Change of the MOS Item Short From Health Survey subscores from baseline to the end of 8 weeks | Baseline and 8 weeks
  The MOS Item Short From Health Survey is a self-report instrument with 36 items, that assesses quality of life through measuring subscales of Physical Function, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Higher subscores indicate better quality of life.
Change in clustering coefficient of brain network from baseline to the end of 8 weeks | Baseline and 8 weeks
  Clustering coefficient is the average of clustering coefficients across all nodes in a network. Higher value indicates greater density and complexity of the entire network.
The change in characteristic path length of brain network from baseline to the end of 8 weeks | Baseline and 8 weeks
  Characteristic path length the average of shortest path length (the minimum number of edges required to connect one node to another node) across any pair of nodes in the network. Lower value indicates higher speed of information transmission in the network.
The change in global efficiency of brain network from baseline to the end of 8 weeks | Baseline and 8 weeks
  Global efficiency is the mean of inverse of the shortest path length between all pairs of nodes in a network. Higher value reflects better functional integration of the network
The change in local efficiency of brain network from baseline to the end of 8 weeks. | Baseline and 8 weeks
  Local efficiency is the mean of the local efficiency across all nodes in whole network. Higher value suggests greater stability of a local network when the local network is interrupted.
The change in normalized clustering coefficient from baseline to the end of 8 weeks. | Baseline and 8 weeks
  Normalized clustering coefficient is the ratio of culstring coefficient of network to the culstring coefficient of random network. Higher value indicates greater local modularization and specialization.
The change in normalized characteristic path length from baseline to the end of 8 weeks | Baselien and 8 weeks
  Normalized characteristic path length is the ratio of characteristic path length of network to characteristic path length of a random network. (the Lp of a random network). Higher value indicates lower global integration effeciency of network.
The change in small-worldness of brain network from baseline to the end of 8 weeks. | Baseline and 8 weeks
  Small-worldness is the ratio of normalized clustering coefficient to normalized characteristic path length. Higher value indicates greater the balance between local specification and global integration of information transmission.
The change in degree centrality of brain network from baseline to the end of 8 weeks | Baseline and 8 weeks
  Degree centrality is the number of direct connections attached to a node. Higher value indicates greater the information transmission between a node and other network nodes.
The change in nodal efficiency of brain network from baseline to the end of 8 weeks | Baseline and 8 weeks
  Nodal efficiency is the average of the inverse of shortest path length between a given node and all other nodes. Higher value indicates greater efficiency of information transmission between a node and other nodes
The change in betweenness centrality of brain network from baseline to the end of 8 weeks | Baseline and 8 weeks
  Betweenness centrality is the number of times a given node lies on one of the paths between all pairs of nodes in a network. Higher value represents greater influence of a node on the overall flow of information in the network.
The change in closeness centrality of brain network from baselien to the end of 8 weeks | Baseline and 8 weeks
  Closeness centrality is the reciprocal of the sum of the shortest path lengths from that node to all other nodes. Higher value reflects greater closeness a node to all other nodes in a network
The change in nodal clustering coefficient of brain network from baseline to the end of 8 weeks | Baseline and8 weeks
  Nodal clustering coefficient is the number of a node's neighbors (nodes directly connecting the node) that are also connected. Higher value indicates greater cliquishness of the subnetwork where the node is located.
The change in nodal local efficiency of brain network from baseline to the end of 8 weeks | Baseline and 8 weeks
  Nodal local efficiency is inverse of shortest path length between all node pairs in the sub-network formed by a given node and its neighbors. Higher value represents greater between the efficiency of information transmission between the node and its neighbors.
The change in nodal shortest path length of brain network from baseline to the end of 8 weeks | Baseline and 8 weeks
  Nodal shortest path length is the average of the shortest path length from a single node to all other nodes in a network. Lower value indicates greater efficiency of information transmission of the node

OTHER OUTCOMES:
The number of participants with treatment-related adverse events recorded in Case Report Form(CRF) at the end of treatment at 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
In order to protect privacy of each participant, there is no plan to share IPD for this study.